CLINICAL TRIAL: NCT01975363
Title: Nanoemulsion Curcumin for Obesity, Inflammation and Breast Cancer Prevention - a Pilot Trial
Brief Title: Pilot Study of Curcumin for Women With Obesity and High Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-13034; NCI-2013-01199 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-08-20; First posted 2013-11-04 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Atypical Ductal Breast Hyperplasia; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ
Keywords: Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Curcumin; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lower dose curcumin) (Experimental): Participants receive 50 mg dose curcumin PO BID for 3 months. Biomarker analyses of breast adipose tissue and plasma samples will be obtained at baseline and 3 months. Breast adipose tissue samples will be obtained via fine needle aspiration. Plasma samples from the baseline blood draw will be assessed for curcumin and also stored at -80°C for biomarker analysis. Assessment of dietary intake by food frequency questionnaires and 24 hour dietary recalls will be used to assess usual dietary habits. All participants will complete a daily log on the date and time of NEC administration, potential adverse events, and medications.
  Interventions: Dietary Supplement: curcumin; Other: Biomarker analysis; Other: Assessment of Dietary Intake; Other: Daily Log
- Arm II (higher dose curcumin) (Experimental): Participants receive 100 mg dose curcumin PO BID for 3 months. Biomarker analyses of breast adipose tissue and plasma samples will be obtained at baseline and 3 months. Breast adipose tissue samples will be obtained via fine needle aspiration. Plasma samples from the baseline blood draw will be assessed for curcumin and also stored at -80°C for biomarker analysis. Asssessment of dietary intake by food frequency questionnaires and 24 hour dietary recalls will be used to assess usual dietary habits. All participants will complete a daily log on the date and time of NEC administration, potential adverse events, and medications.
  Interventions: Dietary Supplement: curcumin; Other: Biomarker analysis; Other: Assessment of Dietary Intake; Other: Daily Log

INTERVENTIONS:
Dietary Supplement: curcumin — Participants will be randomized to either 50 mg BID or 100 mg BID NEC for a 3 month treatment period.
  Other Names: C.I. 75300; C.I. Natural Yellow 3; CU; Diferuloylmethane; NEC
Other: Biomarker analysis — Breast adipose tissue and plasma samples will be obtained at baseline and 3 months for biomarker analyses. Breast adipose tissue samples will be obtained via fine needle aspiration. Plasma samples from the baseline blood draw will be assessed for curcumin/COG and also stored at -80°C for biomarker analyses.
  Other Names: Correlative studies; Breast adipose tissue; plasma samples
Other: Assessment of Dietary Intake — Food frequency questionnaires will be obtained at 0 months and 24-hour dietary recalls will be obtained at 1, 2 and 3 months of the study.
  Other Names: questionnaires
Other: Daily Log — All participants will complete a daily log on the date and time of NEC administration, potential adverse events, and medications.

SUMMARY:
This randomized pilot clinical trial studies a nanoemulsion formulation of curcumin in reducing inflammatory changes in breast tissue in obese women at high risk for breast cancer. Curcumin may reduce inflammation in breast tissue and fat. This may affect the risk of developing breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

i.) To determine whether nanoemulsion curcumnin modulates pro-inflammatory biomarkers in plasma and breast adipose tissue.

SECONDARY OBJECTIVES include:

ii.) To determine the adherence, tolerability and safety of two doses of nanoemulsion curcumin (NEC) in women at high risk for developing breast cancer;

iii.) Evaluate possible correlations between physical factors such as body mass index (BMI), dietary intake and pro-inflammatory effects in plasma and breast adipose tissue.

iv.) Explore additional biomarkers as surrogate endpoints to measure effects of NEC.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive lower dose of nanoemulsion curcumin orally (PO) twice daily (BID) for 3 months.

ARM II: Participants receive 100 mg of nanoemulsion curcumin PO BID for 3 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* Increased risk for breast cancer based on family history, personal history
* Normal mammogram, clinical breast examination in the past 12 months
* >1 year from pregnancy, lactation or chemotherapy
* Body mass index (BMI) between 25 - 40

EXCLUSION CRITERIA:

* Concurrent malignancy or metastatic malignancy of any kind
* Ongoing chemotherapy, radiation therapy, or other cancer-related treatment
* History of a bleeding tendency or current use of Coumadin or other anticoagulants
* Current or previous history of liver, gastrointestinal, hematopoietic, cardiac or renal disease, viral, bacterial, atypical or fungal infections of any organ system and human immunodeficiency virus (HIV) infection
* Pregnant or lactating women
* Concurrent use of hormonal contraception or hormone replacement therapy
* Concurrent use of immunosuppressant medications
* Concurrent use of medications known to inhibit or induce hepatic enzyme cytochrome P450 (CYP) 3A4
* Barriers to fine needle aspiration sampling of breast adipose, including breast implants, history of radiation to both breasts, bilateral mastectomies, and/or insufficient breast adipose tissue for adequate fine needle aspiration (FNA) sampling
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypertension, or psychiatric illness/social situation that would limit compliance with study requirements
* Chronic use of any herbal or dietary supplement containing curcumin or curcuminoids within the 3 months prior to entry on the study or any other supplements that might interact with NEC
* Known sensitivity or allergy to turmeric spices or curry
* Dietary intake of large amounts of curry, turmeric spices or black pepper on a regular basis
* Subjects on a standing regimen of full dose aspirin (>= 325 mg/day), non-steroidal anti-inflammatory drug (NSAID)s or NSAID-containing products

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
Determine the adherence, tolerability and safety of two doses of nanoemulsion curcumin (NEC)in women at high risk for developing breast cancer. | Up to 3 months
  Confidence interval estimates will be obtained from the repeated analysis of variance and two-sample t tests.

SECONDARY OUTCOMES:
Evaluate possible correlations between physical factors such as body mass (BMI), dietary intake and pro-inflammatory effects in plasma and breast adipose tissue. | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu